CLINICAL TRIAL: NCT04895930
Title: A Multi-center, One-arm Clinical Trial of Furmonertinib Combined With Anlotinib as the First-line Treatment in Patients With EGFR Mutation-positive Locally Advanced or Metastatic NSCLC.
Brief Title: Furmonertinib Combined With Anlotinib as the First-line Treatment in Patients With EGFR Mutation-positive NSCLC
Acronym: FOCUS-A
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Baohui Han, Director of department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST-PMR2002
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: EGFR mutations; furmonertinib; anlotinib; non-squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib Plus Anlotinib (Experimental): Furmonertinib (80mg) plus Anlotinib (10mg)
  Interventions: Drug: Furmonertinib; Drug: Anlotinib

INTERVENTIONS:
Drug: Furmonertinib — 80mg/day orally on a continuous dosing schedule. If subjects suffer from AEs, they can get declined dosage (40mg).
  Other Names: AST2818
Drug: Anlotinib — 10mg/day orally from day 1 to 14 of a 21-day cycle. If subjects suffer from AEs, they can get declined dosage (8mg).

SUMMARY:
The aim of this phase Ⅱ study is to evaluate the efficacy and safety of Furmonertinib combined with Anlotinib as the first-line treatment in locally advanced or metastatic non-small cell lung cancer with sensitive EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have voluntarily participated, signed and dated informed consent;
2. Male or female subjects aged ≥18 and ≤75 years old;
3. Locally advanced or metastatic adenocarcinoma NSCLC confirmed by histology or cytology (according to the 8th Edition of the AJCC Staging system), not suitable for surgery or radiotherapy;
4. ECOG score 0-1, and life expectancy no less than 12 weeks according to the investigator's assessment;
5. The tumour harbours one of the most common EGFR mutations (19del or L858R) ;
6. According to RECIST 1.1, subjects have at least one measurable tumor lesion at baseline, and had not received radiotherapy previously;
7. No previous systemic anti-tumor therapy for locally advanced or metastatic NSCLC. For recurrent disease, adjuvant therapy or neoadjuvant therapy may be accepted, but recurrence occurs ≥6 months from stopping treatment;
8. Subjects with stable clinical symptoms of pleural effusion or ascites after symptomatic treatment;
9. For premenopausal women with fertility, the result of serum or urine pregnancy test should be negative within 7 days before the first dose.

Exclusion Criteria:

1. Not lung adenocarcinoma, including lung squamous carcinoma, or mixed histology, etc;
2. Subjects are expected to participate in other clinical studies during this trial period;
3. Imaging evidence showed that the tumor had invaded critical blood vessels;
4. Subjects who receive systemic anti-tumor therapy used for locally advanced or metastatic NSCLC previously;
5. With other malignant tumors at present or history of other malignant tumors within 5 years;
6. Leptomeningeal metastases or central nervous system metastasis requiring emergency treatment;
7. At the beginning of study treatment, any unresolved toxic reaction to prior treatment (e.g., adjuvant chemotherapy) exceeds CTCAE Grade 1;
8. History of ILD, drug-induced ILD, radiation pneumonitis which require steroid treatment, or with suspected clinical manifestations of ILD or high risk factors;
9. Severe gastrointestinal dysfunction may affect the intake, transport or absorption of the study drugs;
10. Recent active digestive diseases or other conditions that may cause gastrointestinal bleeding or perforation;
11. Presence of bleeding constitution or active bleeding; any bleeding event ≥CTCAE grade 3, unhealed wounds, ulcers, or fractures occurred within 28 days prior to the first dose;
12. Any of the following organ function criteria is met (no blood or blood product transfusions, no hematopoietic stimulating factors, no albumin or blood product transfusions within 7 days prior to examination): Absolute value of neutrophil (NE)<1.5 × 109/L, platelet (PLT) count<90 × 109/L, hemoglobin (HGB)<90 g/L; Serum total bilirubin (TBIL)>1.5 × ULN, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>2.5 × ULN (for liver metastases or Gilbert Syndrome, TBIL>3 × ULN, and AST and/or ALT>5 × ULN); Serum creatinine (SCr)>1.5 × ULN, or creatinine clearance<60ml/min. (According to the Cockcroft and Gault formula); Urinary protein ≥ ++, or 24-hour urine protein>1.0g; International normalized ratio（INR）>1.5 and activated partial thromboplastin time (APTT)>1.5 ULN; Fasting blood glucose >10mmol/L；
13. Any of the following cardiac criteria is met：

    * At rest, the mean corrected QT interval (QTc) by ECG > 470 msec；
    * Seriously abnormal of heart rhythm, conduction, or morphology of resting ECG;
    * Any factors that may increase the risk of prolonged QTc or risk of arrhythmic events;
    * Left ventricular ejection fraction (LVEF) < 50%;
    * Uncontrollable hypertension (systolic blood pressure≥150 mmHg and/or diastolic blood pressure≥100 mmHg);
14. With active infection diseases, such as HBV, HCV and HIV;
15. Known or suspected to be allergic to Furmonertinib and Anlotinib and / or other components of their preparations;
16. Pregnancy or lactation;
17. Subjects who are considered ineligible for the study for other reasons according to the investigator's assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 3 years following the first dose of study drugs
  Proportion of subjects whose tumors were assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Approximately 3 years following the first dose of study drugs
  Proportion of subjects whose tumors were assessed as CR, PR or stable disease (SD) according to RECIST 1.1.
Duration of Response (DOR) | Approximately 3 years following the first dose of study drugs
  The time from objective tumor remission (CR or PR) to the progression of the disease or death for any reason.
Disease progression free survival (PFS) | Approximately 3 years following the first dose of study drugs
  The time from the first does of the study drugs to the progression of the disease or death for any reason.
Adverse Events | Until 30 days from the last dose of study drugs or initiation of a new anticancer treatment
  Number of participants with adverse events as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Shi Y, Hu X, Zhang S, Lv D, Wu L, Yu Q, Zhang Y, Liu L, Wang X, Cheng Y, Ma Z, Niu H, Wang D, Feng J, Huang C, Liu C, Zhao H, Li J, Zhang X, Jiang Y, Gu C. Efficacy, safety, and genetic analysis of furmonertinib (AST2818) in patients with EGFR T790M mutated non-small-cell lung cancer: a phase 2b, multicentre, single-arm, open-label study. Lancet Respir Med. 2021 Aug;9(8):829-839. doi: 10.1016/S2213-2600(20)30455-0. Epub 2021 Mar 26. PMID 33780662